CLINICAL TRIAL: NCT04826185
Title: A Randomized, Double-Blinded, Placebo-Controlled Study to Evaluate the Safety, Tolerability, and Efficacy of IMB-1018972 in Patients With Non-obstructive Hypertrophic Cardiomyopathy
Brief Title: A Study to Evaluate the Safety, Tolerability, and Efficacy of IMB-1018972 in Patients With Non-obstructive Hypertrophic Cardiomyopathy Trial
Acronym: IMPROVE-HCM
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Imbria Pharmaceuticals, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: IMB101-007
Record Dates: First submitted 2021-03-18; First posted 2021-04-01 (Actual); Last update posted 2024-04-23 (Actual); Status verified 2024-04

CONDITIONS: Non-obstructive Hypertrophic Cardiomyopathy

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- IMB-1018972 200mg (Experimental)
  Interventions: Drug: IMB-1018972
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: IMB-1018972 — Modified release (MR) oral tablet
  Arms: IMB-1018972 200mg
Drug: Placebo — Matching oral tablet
  Arms: Placebo

SUMMARY:
The purpose of this study is to assess the safety, tolerability, and potential efficacy of IMB-1018972 in patients with non-obstructive HCM.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of Hypertrophic Cardiomyopathy consistent with current US and European guidelines
* Ability to perform an upright treadmill cardiopulmonary exercise test
* Agreement to abide by contraceptive requirements

Exclusion Criteria:

* Clinically significant concurrent condition which could prevent the patient from performing any of the protocol-specified assessments, represent a safety concern if the patient participates in the trial or could confound trial assessments of safety or tolerability
* Women who are pregnant, planning to become pregnant or lactating
* Participation in another clinical study involving a test product or invasive medical device within 28 days (or within 5 elimination half-lives of the respective test product, whichever is longer), prior to first dosing

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 67 (Actual)
Dates: Start 2021-06-14 (Actual); Primary Completion 2023-09-18 (Actual); Study Completion 2023-09-18 (Actual)

PRIMARY OUTCOMES:
Safety and tolerability of IMB-1018972 as measured by incidence and severity of treatment emergent AEs (including AEs leading to study drug discontinuation and AEs leading to death), as well as incidence of treatment emergent SAEs | Baseline through Week 14 Safety Follow-up

SECONDARY OUTCOMES:
Change from baseline of peak oxygen consumption (VO2) and Oxygen uptake efficiency slope (OUES), measured by standardized cardiopulmonary exercise testing (CPET) | Baseline, Week 12

CONTACTS AND LOCATIONS:
Overall Officials: Medical Monitor, Study Chair — Imbria Pharmaceuticals, Inc.
Locations (14):
- United States (13):
  - Imbria Investigational Site, La Jolla, California
  - Imbria Investigational Site, Los Angeles, California
  - Imbria Investigational Site, San Francisco, California
  - Imbria Investigational Site, Chicago, Illinois
  - Imbria Investigational Site, Boston, Massachusetts
  - Imbria Investigational Site, Burlington, Massachusetts
  - Imbria Investigational Site, St Louis, Missouri
  - Imbria Investigational Site, Morristown, New Jersey
  - Imbria Investigational Site, New York, New York
  - Imbria Investigational Site, Charlotte, North Carolina
  - Imbria Investigational Site, Portland, Oregon
  - Imbria Investigational Site, Houston, Texas
  - Imbria Investigational Site, Salt Lake City, Utah
- Imbria Investigational Site, Oxford, United Kingdom

IPD SHARING:
Plan to Share IPD: Undecided